CLINICAL TRIAL: NCT06956859
Title: The Effect of Paternal Skin-to-Skin Contact on Neonatal Physiological Parameters, Comfort and Cortisol Level
Brief Title: The Effect of Paternal Skin-to-Skin Contact on Neonatal Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Associate professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SaglikBilimleri
Record Dates: First submitted 2023-06-23; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Skin to Skin Contact; Newborn; Vitality
Keywords: Skin to skin contact; cortisol; Comfort; newborn; paternalty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin to skin (Experimental): Paternal skin to skin applied to newborns.
  Interventions: Behavioral: Paternal Skin to skin applicated to newborns
- Control Group (No Intervention): Routine maintenance practices were performed in the control group.

INTERVENTIONS:
Behavioral: Paternal Skin to skin applicated to newborns — Paternal Skin to skin applicated to newbornsin the intervention group for 45 minutes. Routine care will be applied to the newborns in the control group. Father Descriptive Information Form, Newborn Descriptive Information Form, Skin-to-Skin Contact Monitoring Form (Newborn/Father), Newborn Comfort
  Arms: Skin to skin

SUMMARY:
This study was planned to examine the effect of skin-to-skin contact between the babies of mothers who gave birth by cesarean section and their fathers on the physiological parameters and comfort of the newborn. The research, which is in a randomized controlled experimental design, will be carried out at the Ministry of Health Sakarya University Training and Research Hospital.

The spouses and babies of 80 pregnant women who were hospitalized with a planned cesarean delivery in Sakarya Training and Research Hospital Gynecology and Child Additional Service Building, will be divided into intervention and control groups by simple randomization method.

Paternal skin-to-skin contact will be applied to newborns in the intervention group for 45 minutes. Routine care will be applied to the newborns in the control group. Father Descriptive Information Form, Newborn Descriptive Information Form, Skin-to-Skin Contact Monitoring Form (Newborn/Father), Newborn Comfort Behavior Scale will be applied to the cases included in the study, body temperature, oxygen saturation, heart rate, respiration will be evaluated, and salivary cortisol analysis will be performed.

The discussion and results of the study will be written in the accompaniment of the findings.

DETAILED DESCRIPTION:
Skin-to-skin contact (TTT) was developed in 1978 in Bogota, Colombia to meet the shortage of incubators required for the care of low-birth-weight babies. It is a method of placement. The sense that occurs in the first seconds after birth in healthy newborns is the sense of touch. Developed countries attach importance to studies that will reveal the effectiveness of this method in order to initiate the parent-newborn relationship and to provide developmental care of the newborn. focused on physiological measures of adaptation to the new environment, such as The results of the study revealed that TTT has many beneficial physiological effects such as increased deep sleep, stable thermoregulation, increased heart rate, respiratory rate and oxygen saturation in newborns. In addition, early skin contact contributes to the development of the nervous system, fewer medical problems, early discharge and reduction in infection rates. Birth is a condition that requires the baby to leave the safe and warm environment in the mother's womb and adapt to a completely foreign environment. It is considered as trauma for the newborn because of its Trauma causes increased stress. Stress negatively affects the evolutionary behavior of newborns and can create intermediate chemicals and hormones in the body that will disrupt the development of the baby. In addition to the immediate negative effects, it can last for the rest of their lives.One of the methods of investigating the degree of stress is to measure the body's cortisol levels; however, it should be noted that stress is not the only cause of the secretion of cortisol into the bloodstream, and other factors such as nutrition, sleep, and sensory simulation can also affect its level. It is known as ". In this case, it can be said that the early postpartum period is critical time to reduce stress. During cesarean section with general / spinal - epidural anesthesia in the operating room, mothers are placed in a supine position, intravenous fluid support is provided, and they are monitored and monitored. Procedures routinely performed on newborn baby after cesarean section; Blood is taken from the umbilical cord of the newborn for the hemogram and blood group, after waiting for 1 minute, the cord is cut and dried and placed under the radiant heater in the operating room. The 1st and 5th minute Apgar scores are evaluated by a midwife who has received NRP training, the choanal and rectal patency is checked, and a mother-baby wristband is put on. The newborn is wrapped in pre-heated operating room covers, and after being shown to the mother for 1-2 minutes, anthropometric measurements (height, body weight, head circumference) are made, vitamin K, hepatitis B vaccine is administered, and the baby is taken to the baby room in the delivery room for the first examination of the baby by the neonatology specialist. . The transfer of the newborn from the delivery room to the room in the gynecology service is provided in approximately 30-50 minutes.

After cesarean births, mother-baby meeting takes place later. This situation negatively affects the comfort of the newborn. Comfort is defined as "an expected result with a complex structure within the physical, psychological, social and environmental integrity of helping individuals related to their needs, obtaining peace and coping with problems". It is often used in babies. The extrauterine environment is an environment where noisy, cool, bright, dry heat and light patterns are not sufficient for newborn babies, unlike intrauterine life, where the baby has difficulty in making movements with the power of gravity. It is said that the practice of TTT with the father during the period until the postpartum routine care of the mother is completed can reduce the problems that the newborn may experience in the early period, provide comfort, and facilitate the adaptation of the father to the new parenting role. It has been determined that they are shorter, they are calmer, and the duration of restlessness is shortened.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for newborns;

* Being born at term (38-42 weeks of gestation)
* Birth weight between 2500-4000gr
* 1st and 5th minute apgar score of 7 and above
* The newborn does not have any health problems
* No surgical intervention

Inclusion criteria for fathers

* No communication problems,
* At least primary school graduate,
* over 18 years old,

Exclusion Criteria:

Neonatal exclusion criteria

* Congenital anomalies
* Metabolic diseases
* Severe periventricular/intraventricular bleeding
* History of minor or major surgery
* Babies from single-parent families
* Babies with intubation and mechanical ventilation
* Having a birth weight of less than 2500 g and more than 4000 g.

Exclusion criteria for fathers

* Unwillingness to participate in the study
* Any contagious disease that can be transmitted through skin contact
* Experiencing fatherhood for the first time
* Not having any contagious disease that can be transmitted through skin contact

Ages: 5 Minutes to 15 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
newborn salivary cortisol level | 0th minute,20th minute,45th minute
  measurement of cortisol in saliva via the cotizol kit
newborn oxygen saturation | 0th minute,20th minute,45th minute
  measurement newborn saturation via pulseoxymeter
newborn body temperature | 0th minute,20th minute,45th minute
  measurement newborn body temperature by thermometer

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Training and Research Hospital, Adapazarı, Sakarya, Turkey (Türkiye)

REFERENCES:
- [Background] Morelius E, Theodorsson E, Nelson N. Salivary cortisol and mood and pain profiles during skin-to-skin care for an unselected group of mothers and infants in neonatal intensive care. Pediatrics. 2005 Nov;116(5):1105-13. doi: 10.1542/peds.2004-2440. PMID 16263996
- [Result] Davis EP, Sandman CA. The timing of prenatal exposure to maternal cortisol and psychosocial stress is associated with human infant cognitive development. Child Dev. 2010 Jan-Feb;81(1):131-48. doi: 10.1111/j.1467-8624.2009.01385.x. PMID 20331658
- [Result] Shonkoff JP, Garner AS; Committee on Psychosocial Aspects of Child and Family Health; Committee on Early Childhood, Adoption, and Dependent Care; Section on Developmental and Behavioral Pediatrics. The lifelong effects of early childhood adversity and toxic stress. Pediatrics. 2012 Jan;129(1):e232-46. doi: 10.1542/peds.2011-2663. Epub 2011 Dec 26. PMID 22201156
- [Result] Takahashi Y, Tamakoshi K, Matsushima M, Kawabe T. Comparison of salivary cortisol, heart rate, and oxygen saturation between early skin-to-skin contact with different initiation and duration times in healthy, full-term infants. Early Hum Dev. 2011 Mar;87(3):151-7. doi: 10.1016/j.earlhumdev.2010.11.012. Epub 2011 Jan 8. PMID 21220191